CLINICAL TRIAL: NCT00455910
Title: Thalidomide for the Treatment of Cytopenias of Patients With Low Risk Myelodysplastic Syndromes
Brief Title: Thalidomide at Low Dose for the Treatment of Patient With Myelodysplastic Syndromes - THAL-SMD-200
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020895; CCPPRB Cochin 2402-1-1928
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: Low risk myelodysplastic syndromes; MDS; Bone marrow diseases; Thalidomide; Cytopenias; Anemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Bone Marrow Diseases; Cytopenia; Anemia | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
The GFM previously conducted a dose-escalating phase II trial of thalidomide in MDS with a minimum dose of 200mg/d and a maximum dose 800mg/d. Responses were evaluated according to IWG criteria at week 16 and thalidomide continued up to week 56 in responders. 82% patients received at least 8 weeks of treatment and were evaluable. 59% had hematological improvement, mainly on the erythroid lineage (Increase of Hemoglobin). Most responses were observed at low doses and between 4 and 8 weeks.

The objectives of this trial (Thal-SMD-20) are to evaluate the efficacy and tolerance of lower doses thalidomide in low risk MDS patients with transfusion-dependant anemia.

DETAILED DESCRIPTION:
Thalidomide:

First part of the trial: 82 patients at 200mg/day given at bedtime x 12 weeks, decreased to 100mg/day if grade 1 or 2 side. Stopped temporally for 1 week if grade 3 or 4 side effects. Then reintroduced at the same dose. If side effects again, definitively stopped.

Responses evaluated at 12 weeks according to IWG criteria for the erythroid lineage

At week 12:

* If no Hematological improvement (HI): increased to 300mg/day for 8 weeks and then eventually to 400mg/day for 8 weeks more, if no HI.
* If Hematological improvement (HI): continued at the same dose.

Second part of the trial: 30 patients treated at 50mg/day x 12 weeks. Responses evaluated at 12 weeks according to IWG criteria for the erythroid lineage

At week 12:

* If no Hematological improvement (HI): increased to 100mg/day for 8 weeks and then eventually to 200mg/day for 8 weeks more, if no HI.
* If Hematological improvement (HI): continued at the same dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years, with IPSS Low or Int-1 MDS
* Transfusion dependant anemia above 2 packed red blood cells (PRBC)/month
* ECOG index = 0, 1, 2
* No peripheral neurological disease

Exclusion Criteria:

* MDS patients with IPSS Int-2 or High
* Patients with less than 2 packed red blood cells (PRBC)/month
* Patients with previous history of venous thrombosis
* Patient treated with EPO +/- G-CSF in the 2 months before inclusion in the protocol
* Patient having received intensive chemotherapy in the 3 months before inclusion in the protocol
* Patient having received Thalidomide in a previous protocol
* Patient presenting an iron, B12 vitamin or folic acid uncorrected deficiency
* Patient with peripheral neurological disease
* Patient not being able to subject itself to a regular clinical and biological follow-up
* Pregnant patient or patient in a period of lactation
* Patient refusing to take a contraceptive treatment through out all the study
* Patient receiving drugs able to interfere with the mechanism of action of Thalidomide
* Patient refusing to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112
Dates: Start 2003-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Efficacy evaluated at week 12 according to the IWG criterias

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Didier Bouscary, MD, Ph-D, Principal Investigator — Groupe Francophone des Myelodysplasies
Locations (20):
- France (20):
  - CHU d'Angers, Angers
  - CH d'Avignon, Avignon
  - CH de la Cote Basque, Bayonne
  - Hopital Avicenne, Bobigny
  - CHU de Brest - Hopital Morvan, Brest
  - CHU Dijon, Dijon
  - CHU Albert Michallon, Grenoble
  - CHRU de Lille - Hopital C. Huriez, Lille
  - CHU de Limoges, Limoges
  - Institut Paoli Calmette, Marseille
  - CHU de Nantes, Nantes
  - CHU de Nice - Hopital de l'Archet 1, Nice
  - Hotel Dieu, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Cochin, Paris
  - Hopital Necker, Paris
  - CH Joffre, Perpignan
  - Centre Henry Becquerel, Rouen
  - CHU Purpan, Toulouse
  - CHU Nancy-Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Bouscary D, Legros L, Tulliez M, Dubois S, Mahe B, Beyne-Rauzy O, Quarre MC, Vassilief D, Varet B, Aouba A, Gardembas M, Giraudier S, Guerci A, Rousselot P, Gaillard F, Moreau A, Rousselet MC, Ifrah N, Fenaux P, Dreyfus F; Groupe Francais des Myelodysplasies (GFM). A non-randomised dose-escalating phase II study of thalidomide for the treatment of patients with low-risk myelodysplastic syndromes: the Thal-SMD-2000 trial of the Groupe Francais des Myelodysplasies. Br J Haematol. 2005 Dec;131(5):609-18. doi: 10.1111/j.1365-2141.2005.05817.x. PMID 16351636
- See also: website of French Group of Myelodysplasia — http://www.gfmgroup.org